CLINICAL TRIAL: NCT02339311
Title: A Home-based Educational Intervention Improves Patient Activation Measures and Diabetes Health Indicators Among Zuni Indians
Brief Title: Zuni Health Initiative - Chronic Disease Education
Acronym: ZHI-CDE
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently entered into the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 10-249
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
Keywords: The study focus is on lifestyle changes and patient activation in diabetic patients by regular monthly visit by the CHRs
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Educational intervention of Lifestyle and patient activation in diabetics — Participants underwent a one hour group didactic session led by Community Health Representatives (CHRs) who subsequently carried out monthly home-based educational interventions to encourage healthy lifestyles, including diet, exercise, and alcohol and cigarette avoidance until follow up at 6 months, when clinical phenotyping and the PAM survey were repeated.

SUMMARY:
One in three people will be diagnosed with diabetes by 2050, and the proportion will likely be higher among Native Americans. Diabetes control is currently suboptimal in underserved populations such as Zuni Indians despite a plethora of new therapies. Patient empowerment is a key determinant of diabetes control, but such empowerment can be difficult to achieve due to resource limitation and cultural, language and health literacy barriers. The investigators will conduct a home-based chronic disease (diabetes) educational intervention using Community Health Representatives (CHRs) to associate improvement in Patient Activation Measures scores (primary outcome) and clinical indicators of diabetes control (secondary outcomes).

DETAILED DESCRIPTION:
The number of American Indians and Alaska Natives (AI/ANs) who have diabetes is growing rapidly, especially among young people. At more than 16%, AI/ANs have the highest age-adjusted prevalence of diabetes among all U.S. racial and ethnic groups [1]. One such population is the Zuni Pueblo home to a small, geographically isolated tribe located in a rural portion of New Mexico, USA. It is home to ~11,000 Zuni Indians and over 90% of all Zunis live in the Pueblo. This socioeconomically disadvantaged population faces a major public health challenge from growing health disparities. Changing lifestyles have led to decreased physical activity and increased caloric intake with high consumption of fast food, soda pop and alcohol. Therefore, the Zuni are experiencing interrelated epidemics of obesity, diabetes, hypertension, kidney disease and intermediate phenotypes.

As part of the Zuni Health Initiative (ZHI), the investigators surveyed participants regarding barriers to healthcare [2], with particular attention to diabetes care. In ZHI the investigators also collected and stored clinical phenotype information and anthropological measurements from all participants. Participants identified the following barriers: access to care, language barriers, limited patient education, and anxiety around diagnosis, fear of chronic disease, reluctance to participate in self-care, resistance to dietary change, and reluctance to engage in regular exercise. The investigators have previously documented suboptimal glycemic control with a high burden of kidney disease among the Zuni [3, 4]. The burden presented by these barriers ultimately translates into a lack of patient activation and engagement in their healthcare, effectively hindering adoption of healthy behaviors. Focus groups subsequently identified common solutions to overcome some of these barriers, including home-based care, point of care testing, individualized exercise and nutrition prescriptions, and care providers with knowledge of the Zuni language, community and culture.

The information gathered during these focus groups [5] is used to design and implement a Zuni culture specific educational intervention in diabetes. The investigators have devised an innovative educational intervention based on the coordination of four key elements: (a) delivering healthcare that incorporated collaborative communication within the healthcare team and emphasized greater autonomy in care, adherence to the medical regimen, and patient-centered goal setting, all while retaining the ability to address the needs of patients, family members, the healthcare team, and/or the healthcare system; (b) providing innovative educational and organizational approaches, as well as behavior change strategies, that enhanced adherence; (c) addressing health beliefs that reduced adherence by over- or under-predicting maladaptive thoughts (e.g., catastrophizing, minimizing, cognitive dissonance, invincibility, or fatalism) or that interfered with weight control; and (d) using technology to address barriers to achieving desired health outcomes.

Sixty participants with type 2 diabetes (T2D) completed a baseline evaluation including physical exam, Point of Care (POC) testing, and the Patient Activation Measure (PAM) survey. Participants then underwent a one hour group didactic session led by Community Health Representatives (CHRs) who subsequently carried out monthly home-based educational interventions to encourage healthy lifestyles, including diet, exercise, and alcohol and cigarette avoidance until follow up at 6 months, when clinical phenotyping and the PAM survey were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes with HbA1c greater than 6.6%
* Zuni Native only
* Age 21-75 yrs
* on diabetes medication

Exclusion Criteria:

* Non-Zuni Native
* Non-diabetic
* Not able to consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is Zuni diabetics with HbA1c level of 6.6% and above in the age range of 21 yrs to 75 yrs old lining in Zuni Pueblo.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Patient Activation | 6 months
  The Patient Activation Measure (PAM) instrument completed by participants using the short form PAM questionnaire [16, 17]. The response options for the 13 questions use a categorical agreement scale with 4 response options: (i) strongly disagree, (ii) disagree, (iii) agree, (iv) strongly agree, and N/A. The raw score is calculated by adding responses to the 13 questions. If all questions are answered (i.e., no "N/A" is used), the range of raw scores would be 13 to 52. If there is at least 1 item with a response of N/A, the total score will be divided by the number of items completed and multiplied by 13 to yield a normalized raw score. All study procedures were repeated 6-months later, following the intervention.

SECONDARY OUTCOMES:
Diabetes associated health indicators | six months
  HbA1c, Glucose, Lipids, BMI

CONTACTS AND LOCATIONS:
Overall Officials: Vallabh Shah, PhD, Principal Investigator — University of New Mexico

REFERENCES:
- [Derived] Shah VO, Carroll C, Mals R, Ghahate D, Bobelu J, Sandy P, Colleran K, Schrader R, Faber T, Burge MR. A Home-Based Educational Intervention Improves Patient Activation Measures and Diabetes Health Indicators among Zuni Indians. PLoS One. 2015 May 8;10(5):e0125820. doi: 10.1371/journal.pone.0125820. eCollection 2015. PMID 25954817